CLINICAL TRIAL: NCT02781051
Title: Increasing Physical Activity Among Breast Cancer Survivors With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122015-072
Record Dates: First submitted 2016-05-03; First posted 2016-05-24 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Depression; Physical Activity; Breast Cancer
MeSH Terms: conditions — Depression; Motor Activity; Breast Neoplasms | interventions — Architectural Accessibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Activity Intervention (Experimental): Participants will participate in a multi-component physical activity intervention for 12 weeks with a 6 month follow up.
  Interventions: Behavioral: Print-based education; Device: Fitbit; Behavioral: Active Living counseling; Other: Facility Access

INTERVENTIONS:
Behavioral: Print-based education — All subjects will be given a copy of Exercise for Health: An Exercise Guide for Breast Cancer Survivors. Topics covered within the book include benefits of exercise in breast cancer survivors; recommendations on type, duration, frequency and intensity of exercise; goal-setting; and advice on overcoming barriers.
Device: Fitbit — Subjects will be provided with a commercially available activity monitor (i.e., Fitbit) and instructed to wear the device daily.
Behavioral: Active Living counseling — The Active Living counseling program consists of 12 weekly group educational sessions, facilitated by project interventionists. These sessions will involve discussion of topics related to increasing physical activity, including: identifying and overcoming barriers, setting goals, and time management.
Other: Facility Access — Subjects will have access to the exercise lab in the UT Southwestern Depression Center consisting of equipment for aerobic exercise (treadmills, stationary bikes, etc.).

SUMMARY:
Pilot study to assess a multi-component intervention to increase physical activity among breast cancer survivors with depression.

DETAILED DESCRIPTION:
The research project is a pilot study to assess the effects of a multi-component intervention in increasing physical activity among breast cancer survivors with depression. Individuals meeting inclusion/exclusion criteria will be enrolled in the 12-week intervention with a 6 month follow up. Intervention components will include print-based education, self-monitoring, Active Living counseling, and facility access. Blood samples will be collected at baseline. Assessments (anxiety, stress, sleep) and sample collection will also occur at 3 time points during the intervention (Weeks 7, 13, and 25). Changes in physical activity will be assessed using Fitbits to measure weekly minutes of moderate/vigorous activity.

ELIGIBILITY:
Inclusion Criteria:

* Positive depression screen (PHQ-9) or current antidepressant treatment
* Report <150 minutes of weekly moderate-to-vigorous physical activity (MVPA) on the GPAQ
* Physically able to engage in physical activity
* Written and verbal fluency in English

Exclusion Criteria:

* Medical condition contraindicating physical activity participation
* Recurrence of breast cancer
* Ductal carcinoma in situ (DCIS) diagnosis
* Cognitively unable to give informed consent
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity Intervention: Participants receive a multi-component physical activity intervention for 12 weeks.
  Print-based education: All subjects will be given a copy of Exercise for Health: An Exercise Guide for Breast Cancer Survivors. Topics covered within the book include benefits of exercise in breast cancer survivors; recommendations on type, duration, frequency and intensity of exercise; goal-setting; and advice on overcoming barriers.
  Fitbit: Subjects were provided with a Fitbit and instructed to wear the device daily.
  Active Living Every Day: 12 weekly group educational sessions, facilitated by project interventionists. Topics included: identifying and overcoming barriers, setting goals, and time management.
  Facility Access: Subjects had access to the exercise lab in the UT Southwestern Depression Center consisting of equipment for aerobic exercise (treadmills, stationary bikes, etc.).
Period: Overall Study
Arm/Group | Physical Activity Intervention
Started | 16
Completed | 14
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Physical Activity Intervention: Participants will participate in a multi-component physical activity intervention for 12 weeks with a 6 month follow up.
  Print-based education: Subjects received the book, Exercise for Health: An Exercise Guide for Breast Cancer Survivors. Topics covered include: benefits of exercise; recommendations on type, duration, frequency and intensity of exercise; goal-setting; and advice on overcoming barriers.
  Fitbit: Subjects were provided a Fitbit and instructed to wear the device daily.
  Active Living counseling: The Active Living counseling program consisted of 12 weekly group educational sessions, facilitated by project interventionists. Discussions will involve topics related to increasing physical activity, such as identifying and overcoming barriers, setting goals, and time management.
  Facility Access: Subjects will have access to the exercise lab in the UT Southwestern Depression Center consisting of equipment for aerobic exercise (treadmills, stationary bikes, etc.).
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.19 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Quick Inventory of Depressive Symptomatology - Self-Rated [Mean (Standard Deviation); unit: units on a scale] — Range: 0-27 Lower scores indicate less depressive symptoms.
  units on a scale | 13.63 (4.5)
Moderate-to-Vigorous Physical Activity [Mean (Standard Deviation); unit: Minutes per week] | 52.4 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Moderate-to-vigorous Physical Activity Measured by Actigraph Accelerometer
Description: Assess changes in physical activity at 6 months following physical activity intervention.
Time Frame: 6 months
Population: 12 participants provided valid baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: minutes per week
Groups:
- Physical Activity Intervention: Participants will participate in a multi-component physical activity intervention for 12 weeks with a 6 month follow up.
  Print-based education: Subjects were given a copy of Exercise for Health: An Exercise Guide for Breast Cancer Survivors. Topics covered within the book include benefits of exercise; recommendations on type, duration, frequency and intensity of exercise; goal-setting; and advice on overcoming barriers.
  Fitbit: Subjects were provided with a Fitbit and instructed to wear the device daily.
  Active Living counseling: The Active Living counseling program consists of 12 weekly group educational sessions. These sessions involved discussion of topics related to increasing physical activity, including: identifying and overcoming barriers, setting goals, and time management.
  Facility Access: Subjects will have access to the exercise lab in the UT Southwestern Depression Center consisting of equipment for aerobic exercise (treadmills, stationary bikes, etc.).
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 12
minutes per week | 56.2 (23.4)

2. Secondary Outcome: Depressive Symptoms Measured by the Quick Inventory of Depressive Symptomatology - Self Report(QIDS-SR)
Description: Assess changes in depressive symptoms at 6 months following physical activity intervention.
  Title: Quick Inventory of Depressive Symptomatology - Self Report(QIDS-SR) Scoring: ranges from 0-27, higher scores indicate more severe symptomatology
Time Frame: 6 months
Population: 14 participants provided follow-up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 14
units on a scale | 9.7 (4.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Physical Activity Intervention
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02781051/Prot_SAP_000.pdf